CLINICAL TRIAL: NCT03678129
Title: Modulation of the Brain Excitatory/Inhibitory (E/I) Balance Through Neuronal Systems in Autism Spectrum Disorder (ASD)
Brief Title: GABA Pathways in Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Grainne McAlonan, Professor, King's College London
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: REC 18/WM/0208
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; E-I balance; AZD7325; pharmacological imaging; GABA
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Clobazam

STUDY DESIGN:
Intervention Model Description: Case-control comparison. Repeated-measures cross-over design. Prepandemic, each subject received each one of the three pharmacological probes in separate visits (i.e., placebo, AZD7325 low dose and AZD7325 high dose), with the order of capsule administration being pseudorandomized. Post pandemic, each participant receives either placebo or 5mg clobazam with the order pseudorandomized.
Who Masked: Participant, Investigator
Masking Description: Participants and investigators are blinded to the drug condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AZD7325 (Other): Prepandemic. Single Dose of Placebo or AZD7325 10mg or AZD7325 20mg random order on visits separated by 1 week
  Interventions: Drug: AZD7325_10; Drug: AZD7325_20; Drug: Placebo
- Clobazam (Other): Post pandemic: Single Dose Placebo or 5mg Clobazam random order on visits separated by 1 week
  Interventions: Drug: Placebo; Drug: Clobazam

INTERVENTIONS:
Drug: AZD7325_10 — Single oral dose (10mg)
  Arms: AZD7325
Drug: AZD7325_20 — Single oral dose (20mg)
  Arms: AZD7325
Drug: Placebo — Single oral dose placebo (capsule)
Drug: Clobazam — Single dose (5mg)
  Arms: Clobazam

SUMMARY:
This study investigates the brain response to a single acute dose of a GABAa receptor acting drug (Benzodiazepine or positive allosteric modulator) compared to a single dose of placebo in adults with and without autism spectrum disorder.

DETAILED DESCRIPTION:
Previous research suggests that GABAergic drug compounds could shift brain excitation and inhibition (E-I) in the healthy brain and in neurodevelopmental psychiatric conditions, such as autism spectrum disorder (ASD) - where this balance is disrupted. A study by Ajram et al. (2017) has shown an E-I shifted towards more GABA in individuals with ASD, and not in controls, after a single dose of the anti-glutamatergic and pro-GABAergic drug Riluzole. Moreover, brain connectivity patterns in ASD patients where shifted towards the ones observed in the control group. However, it was unclear whether this changes could be driven by GABA receptors, thus more specific probes may help to clarify the mechanism underlying the E-I coordination in ASD. Therefore, this study will use neuroimaging and electrophysiology to investigate the brain E-I coordination in ASD compared to control participants when the system is responding to a single dose of a GABA-A acting drug.

Please note, when first registered we had access to the specific GABA-A (AZD7325) receptor positive allosteric modulator. Following a pause in the study over the Covid pandemic this compound was not longer available. Therefore, we have updated the protocol and instead are using clobazam, a GABA-A/benzodiazepine receptor agonist. We have also now expanded the information about measures acquired in this study.

Up to 50 adult individuals with ASD and 50 neurotypical adults (25 males and 25 females per group) will be invited to participate. Prior to the pandemic, each participant received a single dose of the drug (10mg or 20mg AZD7325) or matched placebo. Following ethics amendment post pandemic, AZD7325 will no longer be used and participants will receive 5mg of clobazam or placebo.

Brain activity and neurochemistry will be investigated using magnetic resonance imaging, EEG and psychophysics. Further data will be collected through questionnaires, behavioural tasks, blood samples, and retinal physiology.

Our study is defined as a Basic Science study in human participants. It does not address safety or clinical efficacy and the UK Medicines and Health Regulatory Authority (MHRA) has confirmed that our protocol is therefore not a clinical trial of an Investigational Medicinal Product (IMP) as defined by the EU Directive 2001/20/EC

ELIGIBILITY:
Inclusion Criteria

For all participants:

1. Calendar age above 18 years.
2. Able to give informed consent.
3. Not pregnant or breastfeeding.
4. Ideally prescription medication free during the 2-week period preceding a study visit. However, occasional use of over-the-counter medication (e.g. painkillers) on an as needed basis (and not on the day of study visit) may be permitted. In addition, regular prescription medication (use of a stable dose over the two months preceding participation) with a drug that does not affect glutamate or GABA directly may be permitted. Also permitted is topical medication without systemic exposure.

For individuals with ASD:

1. Diagnosis of ASD confirmed on the Autism Diagnostic Interview-Revised (ADI-R) if a relative is available and/or on the Autism Diagnostic Observation Schedule (ADOS-2).

For all relatives:

1. Aged under 18 years.
2. Does not know the participant personally at present or in their childhood.

Exclusion Criteria:

For all participants

1. History of allergy/idiosyncrasy to AZD7325 or chemically related compounds or excipients which may be employed in the study or to any other drug used in the past.
2. Subject has taken systemically (po, iv) any potent or moderate CYP3A4 or CYP2C9 inhibitor or inducer, 1 month prior to screening (topical or inhaled are permitted) such as: aprepitant, barbiturates, carbamazepine, clarithromycin, erythromycin, cyclosporine, diltiazem, efavirenz, fluconazole, HIV protease inhibitors, glucocorticoids, itraconazole (oral/IV), ketoconazole, nefazodone, nevirapine, phenytoin, pioglitazone, primidone, rifabutin, rifampicin, telithromycin, St. John's wort, verapamil.
3. Clinically relevant history or presence of any medical disorder, potentially interfering with this study.
4. Clinically relevant abnormality at screening as judged by the investigator.
5. History of or current abuse of drugs (including prescription medication) or alcohol or solvents.
6. Participation in a research study involving a pharmacological probe or drug trial within last month or more than four in the previous 12 months
7. Subjects with a history of epilepsy, seizures or episodes of unexplained and unprovoked loss of consciousness.
8. Anyone with a history or examination which indicates laboratory testing is needed will be excluded from the study.
9. Intelligence Quotient below 70.

Reproductive safety: Male study participants who are sexually active should avoid procreation for 1 week after study drug administration. Avoidance of procreation can be through use of a highly effective contraception method by the study participant or by the partner. In this case, effective means of contraception are defined as tubal occlusion, copper banded intrauterine device, levonorgestrel medicated intra uterine system (e.g., Mirena), medroxyprogesterone injections (e.g. Depo-Provera), etonogestrel implants (e.g., Implanon, Norplan), normal and low dose combined oral contraceptive pills, norelgestromin / EE transdermal system, intravaginal device (e.g., EE and etonogestrel) and desogestrel (Cerazette).

Pregnancy or breastfeeding (is a routine exclusion for research MRI scanning). Female study participants must be willing to use one form of highly effective non-hormonal contraception for one week after study drug administration. This would include a vasectomised partner (sole partner), tubal occlusion, intrauterine system [IUS]/hormonal coil or copper containing intrauterine device or copper containing IUD, or true abstinence (when this is in line with the preferred and usual lifestyle of the subject). Women should have been stable on their chosen method of birth control for a minimum of 2 months before entering the study. Participants must agree to undergo a pregnancy test prior to each administration of study drug.

For individuals with ASD:

1. ASD caused by a known genetic syndrome, e.g. Fragile X, 22q11 deletion syndrome.
2. Currently treated for epilepsy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Brain activation and connectivity response to GABAergic stimulation as assessed by functional magnetic resonance imaging. | Data collected on up to 3 visit days per participant. Completed within up to 1 year.
  Comparing whole brain blood-oxygen-level-dependent (BOLD) activation (institutional units) during the resting state in cases and controls when a single oral dose of GABA-A receptor acting compound administered versus the placebo condition.
Brain electrophysiological activity task-free electroencephalography (EEG) | Data collected on up to 3 visit days per participant. Completed within up to 1 year
  Case-control comparison of task-free Electroencephalogram (EEG) during placebo and when GABA-A compound administered. Analyses approaches will include examining power and phase information across different frequencies and aperiodic signal analysis (1/f like); and evaluation of power spectrum and functional connectivity across source localisations.
Brain oscillations under sensory stimulation | Data collected on up to 3 visit days per participant. Completed within up to 1 year
  Brain oscillations (spectral perturbations) and event-related potentials will be recorded during sensory stimulation - auditory (odd-ball) and visual (contrast saturation, face perception/N170) tasks using electroencephalography during placebo and when GABA-A compound administered.

OTHER OUTCOMES:
Brain excitation and inhibition response to GABAergic stimulation as assessed by magnetic resonance spectroscopy. | Data collected on up to 3 visit days per participant. Completed within up to 1 year
  Quantification and case-control comparison of brain metabolites relevant to regulation of excitation and inhibition (focus on Glx, GABA, GSH) using proton magnetic resonance spectroscopy when 'at rest' (placebo) and when activated by GABA-A compound.
Tactile perception | Data collected on up to 3 visit days per participant. Completed within up to 1 year
  Case-control comparison of tactile discrimination during placebo and when GABA-A compound administered.
Electroretinogram | Data collected on up to 3 visit days per participant. Completed within up to 1 year
  Case-control comparison of ERG acquired with hand held device during placebo and when GABA-A compound administered. three stimulus protocols: i) the standard white flash; ii) the standard 30-Hz flickering protocol; iii) the photonic negative response (PhNR) protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Grainne McAlonan, PhD, Principal Investigator — King's College London, UK
Locations (1):
- King's College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No